CLINICAL TRIAL: NCT04702958
Title: Mechanistic Insights From Longitudinal Changes in Blood and Urine Proteins to Explain Efficacy and Safety of Torsemide vs Furosemide After a Heart Failure Hospitalization
Brief Title: TRANSFORM-HF Ancillary Mechanistic Study
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Duke University (Other); George Mason University (Other); University of Maryland, Baltimore (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01HL154768-01 (NIH); R01HL154768-01 (NIH)
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Single biomarkers: high sensitive cardiac troponin T (hs-cTnT), amino terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor 15 (GDF-15), Cystatin C, high sensitive C-reactive protein (hsCRP), and interleukin 6 (IL6).
  * Urinary biomarkers: albumin, beta-2 microglobulin (B2M), cystatin C, epidermal growth factor (EGF), neutrophil gelatinase-associated lipocalin (NGAL/Lipocalin-2), osteopontin (OPN), uromodulin (UMOD)
  * Targeted discovery proteomics: Olink CARDIOVASCULAR III (CVD III) panel
  * Covid-19 antibodies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Torsemide: Patients enrolled in the TRANSFORM-HF study randomized to Torsemide, or patients prescribed Torsemide at hospital discharge
- Furosemide: Patients enrolled in the TRANSFORM-HF study randomized to Furosemide, or patients prescribed Furosemide at hospital discharge

SUMMARY:
Patients with heart failure are frequently treated with diuretics, including furosemide and torsemide, but it is not known if one is better than the other. The TRANSFORM-HF trial is studying if torsemide is superior than furosemide for reducing the endpoint of death or hospitalization, but is not designed to study why. This ancillary study seeks to measure proteins in the blood and urine to help explain the underlying mechanism for why patients who take one of these diuretics may have better outcomes than patients who take the other.

DETAILED DESCRIPTION:
Patients who are enrolling in the TRANSFORM-HF study or being prescribed Torsemide or Furosemide at hospital discharge will provide blood and urine at the time of study enrollment (within 72 hours of hospital discharge) and at 90 days (+/- one week) after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the TRANSFORM-HF trial or prescription of Torsemide or Furosemide
* Willing to provide blood and urine sample at enrollment and follow-up

Exclusion Criteria:

* Inability or unwillingness to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll a subset of patients who are enrolling in the TRANSFORM-HF study during a hospitalization for acute HF, or who are prescribed Torsemide or Furosemide at hospital discharge, and who are willing to provide biospecimens for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Differences in proteomic protein clusters between treatment groups | baseline
  How the biomarkers are different between groups
Differences in trajectories of protein clusters between treatment groups | 90 days
  How the protein clusters change over time from baseline to 90 days

SECONDARY OUTCOMES:
Differences in single biomarkers and biomarker trajectories between treatment groups | baseline and 90 days
  How the biomarkers are different between groups at baseline and how the biomarkers change over time from baseline to 90 days
Differences in urinary protein levels between treatment groups | baseline
  How the in urinary protein levels are different between patient prescribed Torsemide vs Furosemide

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Cooper, MD, MHS, Principal Investigator — Northwell Health; Christopher deFilippi, MD, Principal Investigator — Inova Health Care Services
Locations (9):
- United States (9):
  - Yale University School of Medicine, New Haven, Connecticut
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Baltimore VA, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Northwell Health, Manhasset, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Inova Health System, Falls Church, Virginia
  - Sentara Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No